CLINICAL TRIAL: NCT01407874
Title: A Randomized, Double-Blind, Dose-Response Study of the Safety and Uric Acid Effects of Oral Ulodesine Added to Allopurinol in Subjects With Gout and Concomitant Moderate Renal Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCX4208-204
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Gout; Hyperuricemia; Arthritis; Joint Disease; Renal Insufficiency
Keywords: Gout; Hyperuricemia; Arthritis; Joint Disease; Allopurinol; Renal Insufficiency
MeSH Terms: conditions — Gout; Hyperuricemia; Arthritis; Joint Diseases; Renal Insufficiency | interventions — ulodesine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): Placebo + Allopurinol 200mg
  Interventions: Drug: Placebo
- Ulodesine (BCX4208) 5mg (Experimental): BCX4208 5mg + Allopurinol 200 mg
  Interventions: Drug: Ulodesine (BCX4208) 5 mg
- Ulodesine (BCX4208) 10mg (Experimental): BCX4208 10mg + Allopurinol 200mg
  Interventions: Drug: Ulodesine (BCX4208) 10 mg

INTERVENTIONS:
Drug: Placebo — Oral dose administered daily for 84 days.
  Arms: Placebo
Drug: Ulodesine (BCX4208) 5 mg — Oral dose administered daily for 84 days.
  Arms: Ulodesine (BCX4208) 5mg
Drug: Ulodesine (BCX4208) 10 mg — Oral dose administered daily for 84 days.
  Arms: Ulodesine (BCX4208) 10mg

SUMMARY:
To evaluate the overall safety and tolerability of ulodesine when combined with allopurinol in subjects with moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to < 70 years
2. Have read and signed the Informed Consent Form
3. Documented diagnosis of gout
4. Documented moderate renal insufficiency
5. Calculated creatinine clearance of ≥ 30 and < 60 mL/min
6. Willing and able to take allopurinol 200 mg every day for the duration of the Treatment
7. Female participants must be sexually abstinent for 4 weeks prior to Day 1 and continue abstinence for 4 weeks after completion of study drug, surgically sterile, postmenopausal,use oral contraceptives for three months prior to study drug dosing through 4 weeks after completion of study drug, an intrauterine device for 8 weeks prior to study drug dosing through 4 weeks after completion of study drug,double barrier contraception method for 4 weeks prior to study drug dosing through 4 weeks after completion of study drug administration
8. Male participants must be sexually abstinent for 4 weeks prior to Day 1 and continue abstinence through 90 days after completion of study drug, be > 1 year postvasectomy, agree to use a condom with spermicide from the start of study drug dosing through 90 days after completion of study drug.
9. Willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act (HIPAA)

Exclusion Criteria:

1. Unable to tolerate allopurinol 200 mg every day
2. Prior randomization in a clinical study with BCX4208
3. Unstable cardiac disease such as: unstable angina, symptomatic arrhythmia, signs or symptoms compatible with NYHA Class III or Class IV functional status for congestive heart failure or angina, history of long QT syndrome, or QTc interval < 350 msec or > 475 msec
4. Poorly controlled hypertension
5. History of severe renal insufficiency
6. Alanine aminotransferase or aspartate aminotransferase values > 2.0 x upper limit of normal
7. CD4+ cell counts by flow cytometry < 500 cells/mm3
8. Hemoglobin < 10 g/dL or > 18 g/dL (males) or < 10 g/dL or > 17 g/dL (females)
9. White blood cell count < 3.7 x 109/L or > 11 x 109/L
10. Female subjects who are pregnant, breastfeeding, or planning a pregnancy within the next 4 months
11. Positive serology for hepatitis B surface antigen or hepatitis C antibody or HIV type 1
12. Immunocompromised due to illness or organ transplant
13. Use of systemic immunosuppressive medications or disease-modifying antirheumatic drugs
14. Use of azathioprine or 6-mercatopurine within 14 days of first dose of allopurinol
15. Use of hydrochlorothiazide in doses > 50 mg per day
16. Planned use of herbal or dietary supplements
17. Recipient of any live or attenuated vaccine within 6 weeks of Screening
18. Planned use of uric acid-lowering drugs other than allopurinol
19. Use of systemic corticosteroids within 4 weeks prior to Day 1
20. Use of any investigational drug within 30 days prior to signing the ICF
21. History of clinically significant and relevant drug allergies
22. History of chronic or recurrent infections
23. History of any type of cancer not successfully treated or in full remission for 12 months prior to Screening
24. History of alcohol or drug abuse within the year prior to the signing of the ICF, or current evidence of substance dependence or abuse
25. Use of other prohibited medications within the timeframes specified in the protocol
26. Other medical conditions which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall safety and tolerability of ulodesine when combined with allopurinol in subjects with moderate renal insufficiency by assessment of percent change from baseline in CD4+ lymphocytes at Day 85. | 85 days
  Level of CD4+ lymphocytes to be measured at Day 85 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Hollister, MD, PhD, Study Director — BioCryst Pharmaceuticals
Locations (10):
- United States (10):
  - Mobile, Alabama
  - Peoria, Arizona
  - Irvine, California
  - Oldsmar, Florida
  - Honolulu, Hawaii
  - Newton, Kansas
  - Knoxville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Alexandria, Virginia